CLINICAL TRIAL: NCT01481688
Title: Intradialytic Exercise for Enhanced Dialysis Adequacy and Solute Removal in Chronic Kidney Disease Patients: A Randomised Controlled Trial.
Brief Title: Enhancing Dialysis Adequacy: Effects of Intradialytic Exercise
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangor University (Other)
Collaborators: Betsi Cadwaladr University Health Board (Other Government); B.Braun Avitum AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11/WA/0112; Kirkman 11/WA/0112 (Other Grant/Funding Number: R & D Reference Number)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Kidney Disease
Keywords: Dialysis adequacy; Urea clearance; Phosphate clearance; Beta 2 microglobulin clearance; Intradialytic exercise; Haemodialysis patients
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Routine haemodialysis sessions as per usual
- Intradialytic exercise (Experimental): One hour of exercise completed during haemodialysis.
  Interventions: Other: Exercise
- Extra time (Active Comparator): 30 minutes extra dialysis time.
  Interventions: Other: Extra time

INTERVENTIONS:
Other: Exercise — Exercise During Dialysis Patients will be asked to carry out cycling exercise for 60 minutes during the third quarter of their routine haemodialysis session. Exercise can be carried out in ten minute bouts with several minutes rest between bouts.
  Arms: Intradialytic exercise
Other: Extra time — An extra 30 minutes will be added to the currently prescribed treatment time of each patient.
  Arms: Extra time

SUMMARY:
The purpose of this study is to investigate whether intradialytic exercise increases removal of waste products from blood, in comparison to the traditional prescription of increasing dialysis duration.

DETAILED DESCRIPTION:
For patients with severe chronic kidney disease, regular dialysis to remove toxins and waste products from the blood is essential to maintain life. The adequacy of dialysis is quantified by the removal of these toxic solutes and is an important parameter in the assessment of the therapy.

Previous efforts to enhance urea clearance have centered around factors such as increasing dialysis dose by increasing dialysis time or carrying out more frequent dialysis sessions. However this concept is confronted with the barriers of patient compliance and cost implications. Many patients are resilient to increasing their dialysis time, presenting a major challenge for enhancing the efficacy of dialysis therapy. Therefore, alternative methods of improving dialysis adequacy, with interventions aimed at enhancing solute clearance, are highly warranted.

One such intervention could be exercising during haemodialysis (HD). 85% of the body is comprised of lean tissue, of which 73% is water. As many toxic solutes are water based, large amounts will be stored in the muscle. When sitting at rest during HD the blood flow to the muscles is four times less compared to the major organs. Additionally, the HD process causes blood vessels to constrict, further restricting blood flow to the muscle. Consequently there is insufficient blood flow to remove the toxins stored in the muscle. By exercising during dialysis, blood flow to the muscle is increased to sustain the demand for oxygen and energy, thereby allowing toxic solutes to be removed and cleared through the dialysis machine.

Therefore the aim of this study is to implement an efficient exercise intervention during dialysis and determine its effects on dialysis adequacy in comparison to the traditional prescription of increased dialysis time. In particular, the study aims to explore the acute effects of exercise during dialysis on the removal of several established uremic toxins.

ELIGIBILITY:
Inclusion Criteria:

* Stage 5 Chronic Kidney Disease
* Receiving maintenance haemodialysis for > 3 months

Exclusion Criteria:

* Unable to give consent
* Present with contraindications to take part in exercise
* Haemoglobin <11 g/dL
* Access recirculation
* Chronic persistent hypotension with pre dialysis systolic blood pressures <100mgHg.
* Episodic treatment induced hypotension with frequent drops in intradialytic systolic blood pressure >30mmgHg
* Unstable medical condition
* Currently taking medication affecting urea or creatinine generation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Urea clearance | One dialysis session
  The primary outcome is urea clearance which will be measured by continuously sampling waste dialysate from an entire dialysis session.

SECONDARY OUTCOMES:
Urea clearance | One dialysis session
  Urea clearance which will be measured by continuously sampling UV absorbance of waste dialysate during an entire dialysis session.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie H Macdonald, PhD, Study Director — Bangor University
Locations (1):
- Renal unit, Ysbyty Gwynedd, Betsi Cadwaladr University Health Board, Bangor, Gwynedd, United Kingdom

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639